CLINICAL TRIAL: NCT04503512
Title: Effect of Excision of the Fat Pad in Total Knee Replacement Surgery. A Randomised Controlled Trial
Brief Title: Surgical Excision of the Fat Pad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4263
Record Dates: First submitted 2019-08-23; First posted 2020-08-07 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-06

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non removal of fat pad (Active Comparator): Non removal of fat pad
  Interventions: Procedure: non removal of fat pad
- Removal of fat pad (Active Comparator): Removal of fat pad
  Interventions: Procedure: removal of fat pad

INTERVENTIONS:
Procedure: removal of fat pad — Removal removal of fat pad
  Arms: Removal of fat pad
Procedure: non removal of fat pad — non removal of fat pad
  Arms: Non removal of fat pad

SUMMARY:
Introduction:

The infrapatellar fat pad (Hoffa's fat pad) is a structure which is located intra-articularly. Its function is not well known. During knee replacement surgery, some surgeons would prefer removing the whole of the fat pad as this can improve exposure of the knee joint, as it can affect exposure of the knee joint which will in turn make the procedure slightly more efficient. Other surgeons would rather resect the minimum amount and preserve the bulk of the structure as anecdotally this is thought to decrease the level of post operative pain. This surgical step fat pad resection is a very small part of the whole total knee replacement procedure.

A previous retrospective review of patients whose fat pad had been removed showed that they were nearly twice as likely to experience postoperative pain (P = 0.0005), while another study showed that they are at a slight risk of patellar tendon shortening.

A randomised controlled trial of 68 patients did not show any difference in patella tendon length at six months and no difference in pain relief in both groups 3. However this study did not evaluate the functional outcome in both groups.

To our knowledge, there are no RCT looking at the effect of the excision or preservation of the fat pad in TKR and the functional outcomes post operatively.

Study Hypothesis:

Excision of Hoffa's fat pad during total knee replacement surgery does not affect functional outcome, pain level after surgery or the patella tendon length at either one or two years.

DETAILED DESCRIPTION:
RCT of excision or preservation of fat pad in TKR and the functional outcomes post operatively

ELIGIBILITY:
Inclusion Criteria:

* 1- Primary total knee replacement for knee osteoarthritis

Exclusion Criteria:

1. Revision Surgery.
2. Primary Knee Replacement for pathologies other than Osteoarthritis.
3. Previous knee fractures around the knee.
4. Previous confirmed intra-articular infections.
5. Non English speaking/reading patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-10-23 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Koos Knee Score | 3 months post op,
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury.

CONTACTS AND LOCATIONS:
Overall Officials: A Howard, Study Director — Liverpool University Hospitals NHS Foundation Trust
Locations (1):
- Broadgreen Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No